CLINICAL TRIAL: NCT01256762
Title: A Randomized Phase II Study Of Imetelstat (GRN163L) In Combination With Paclitaxel (With Or Without Bevacizumab) in Patients With Locally Recurrent Or Metastatic Breast Cancer
Brief Title: Imetelstat in Combination With Paclitaxel (With or Without Bevacizumab) in Patients With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP14B014
Record Dates: First submitted 2010-12-02; First posted 2010-12-09 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-12

CONDITIONS: Locally Recurrent or Metastatic Breast Cancer
Keywords: imetelstat; imetelstat sodium; GRN163L; telomerase inhibitor; telomerase inhibition; metastatic breast cancer; locally recurrent breast cancer; Bevacizumab; Paclitaxel; Avastin; Taxol; HER-2-negative; First-Line Chemotherapy; Second-Line Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — imetelstat; GRN163L peptide; Bevacizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imetelstat + Paclitaxel (with or without bevacizumab) (Experimental)
  Interventions: Drug: Imetelstat sodium; Drug: Bevacizumab; Drug: Paclitaxel
- Paclitaxel (with or without bevacizumab) alone (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Imetelstat sodium — Imetelstat is administered at a dose of 300 mg/m2 on day one of a 21 day cycle.
  Other Names: GRN163L
  Arms: Imetelstat + Paclitaxel (with or without bevacizumab)
Drug: Bevacizumab — Bevacizumab is administered at 15 mg/kg on day one of a 21 day cycle
  Other Names: Avastin
Drug: Paclitaxel — Paclitaxel is administered at 90 mg/m2 on days one and eight of a 21 day cycle
  Other Names: Taxol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of treatment with imetelstat + paclitaxel (with or without bevacizumab) versus paclitaxel (with or without bevacizumab) alone for patients with locally recurrent or metastatic breast cancer who have not received chemotherapy or have received one non-taxane based chemotherapy for metastatic breast cancer.

DETAILED DESCRIPTION:
Patients will be randomized in a 1:1 ratio to imetelstat + paclitaxel (with or without bevacizumab) versus paclitaxel (with or without bevacizumab) alone.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed adenocarcinoma of the breast that is either locally recurrent or metastatic. Locally recurrent disease must not be amenable to surgical resection or radiation with curative intent
* Either have not received chemotherapy or may have had one prior non-taxane chemotherapy regimen for metastatic disease (there are no restrictions on prior hormonal therapy)
* Prior use of bevacizumab is allowed provided that it was not administered in combination with a taxane
* ECOG performance status 0-1
* Adequate bone marrow reserve as indicated by:

  * ANC > 1500/uL (without use of growth factors within 7 days)
  * Platelet count > 100,000 (without transfusion in prior 7 days)
  * Hemoglobin > 9.0 g/dL

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Locally recurrent disease amenable to resection with curative intent
* HER-2-positive breast cancer
* Active central nervous system (CNS) metastatic disease including those patients receiving radiotherapy and/or steroid treatment (within the last 3 months)
* Prior adjuvant or neoadjuvant taxane chemotherapy within 12 months prior of first relapse
* Investigational therapy within 4 weeks of first study drug administration
* Prior radiation, cytotoxic, or hormonal therapy within 2 weeks of first study drug administration
* Therapeutic anti-coagulation or regular use of anti-platelet therapy within 2 weeks prior to first study drug administration (low dose anti-coagulant therapy to maintain patency of a vascular access device is allowed)
* Grade ≥ 2 neuropathy
* Uncontrolled clinically significant atrial or ventricular arrhythmias (unless pacemaker in place)
* Severe conduction disturbance including clinically significant QTC prolongation > 450 ms (unless pacemaker in place)
* Active or chronically recurrent bleeding (e.g., active peptic ulcer disease)
* Clinically relevant active infection
* Known positive serology for human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Occurring post randomization through end of study period (9 mos. after the last participant is randomized)
  Defined as the time from randomization to documented disease progression, as determined by the investigator's assessment according to RECIST, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective response | Occurring post randomization through end of study period (9 mos. after the last participant is randomized)
  Objective response as determined by the investigator according to RECIST for patients with measurable disease at baseline.
Clinical benefit rate | Occurring post randomization through end of study period (9 mos. after the last participant is randomized)
  Clinical response rate includes patients with objective response and stable disease lasting at least 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ted Shih, PharmD, Study Director — Geron Corporation; Kathy Miller, MD, Principal Investigator — Indiana University School of Medicine
Locations (55):
- United States (50):
  - Clearview Cancer Center, Huntsville, Alabama
  - Alta Bates Summit Medical Center, Berkeley, California
  - Southbay Oncology Hematology Partners, Campbell, California
  - Cancer Care Associates, Fresno, California
  - Memorial Miller Hospital, Long Beach, California
  - St. Joseph Hospital, Orange, California
  - Desert Regional Comprehensive Cancer Center, Palm Springs, California
  - UC San Diego, San Diego, California
  - Redwood Regional Medical Group, Santa Rosa, California
  - Univ. Colorado at Denver, Aurora, Colorado
  - Connecticut Oncology & Hematology, Torrington, Connecticut
  - Medical Oncology Hematology, Waterbury, Connecticut
  - Florida Oncology Associates, Jacksonville, Florida
  - Hematology Oncology Associates, Port Saint Lucie, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northeast Georgia Cancer Care, Athens, Georgia
  - Peachtree Hematology Oncology, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - Kootenai Medical Center, Post Falls, Idaho
  - Ingalls Memorial Hospital, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - Mid Illinois Hematology & Oncology, Normal, Illinois
  - Cancer Treatment Centers of America, Zion, Illinois
  - Indiana University, Indianapolis, Indiana
  - Community Hospitals of Indiana, Indianapolis, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Montgomery Cancer Care, Mount Sterling, Kentucky
  - Michigan State University, East Lansing, Michigan
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Prohealth Associates, Lake Success, New York
  - Stony Brook University, Stony Brook, New York
  - Carolinas Hematology/Oncology, Charlotte, North Carolina
  - Moses Cone Medical System, Greensboro, North Carolina
  - Case Western Reserve Univ., Cleveland, Ohio
  - Mercy Physicians of Oklahoma, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Kaiser Northwest, Portland, Oregon
  - Pinnacle Health, Harrisburg, Pennsylvania
  - Penn. State Univ., Hershey, Pennsylvania
  - The Jones Clinic, Germantown, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Scott & White Healthcare, Temple, Texas
  - Northern Utah Associates, Ogden, Utah
  - Peninsula Cancer Institute, Newport News, Virginia
  - Medical Oncology Associates, Spokane, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Canada (5):
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - Stronach Regional Cancer Centre at Southlake, Newmarket, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Services Centre, Toronto, Ontario
  - McGill University, Montreal, Quebec

REFERENCES:
- [Background] Hochreiter AE, Xiao H, Goldblatt EM, Gryaznov SM, Miller KD, Badve S, Sledge GW, Herbert BS. Telomerase template antagonist GRN163L disrupts telomere maintenance, tumor growth, and metastasis of breast cancer. Clin Cancer Res. 2006 May 15;12(10):3184-92. doi: 10.1158/1078-0432.CCR-05-2760. PMID 16707619
- [Background] Goldblatt EM, Gentry ER, Fox MJ, Gryaznov SM, Shen C, Herbert BS. The telomerase template antagonist GRN163L alters MDA-MB-231 breast cancer cell morphology, inhibits growth, and augments the effects of paclitaxel. Mol Cancer Ther. 2009 Jul;8(7):2027-35. doi: 10.1158/1535-7163.MCT-08-1188. Epub 2009 Jun 9. PMID 19509275
- [Background] Herbert BS, Wright WE, Shay JW. Telomerase and breast cancer. Breast Cancer Res. 2001;3(3):146-9. doi: 10.1186/bcr288. Epub 2001 Feb 22. PMID 11305948